CLINICAL TRIAL: NCT04406194
Title: Open-label,Randomised,Single Oral Dose,Two-period,Cross-over Trial to Assess to Bioequivalence of Favicovir 200 mg FT in Comparison With Avigan 200 mg FT in Healthy Male Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Favipiravir 200 mg Film Tablet (ATABAY, Turkey) Under Fasting Conditions
Acronym: Favipiravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atabay Kimya Sanayi Ticaret A.S. (Industry)
Collaborators: Novagenix Bioanalytical Drug R&D Center (Network); Farmagen Ar-Ge Biyot. Ltd. Sti (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NOV2020/1917
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Bioequivalence
Keywords: COVID-19 drug treatment; Antiviral Agents; Favipiravir; Novagenix; Farmagen
MeSH Terms: interventions — Motion Pictures; favipiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAVICOVIR then AVIGAN (Experimental): Participants first received Favicovir 200 mg FT manufactured by Atabay in a fasting state. After a washout period of 48 hours, they then received Avigan FT200 mg manufactured by Toyama Chemical Industry Co.Ltd./Japan in a fasting state.
  Interventions: Drug: FAVICOVIR 200 mg Film Tablet; Drug: AVIGAN 200 mg Film Tablets
- AVIGAN then FAVICOVIR (Experimental): Participants first received Avigan FT200 mg manufactured by Toyama Chemical Industry Co.Ltd./Japan in a fasting state. After a washout period of 48 hours, they then received Favicovir 200 mg FT manufactured by Atabay in a fasting state.
  Interventions: Drug: FAVICOVIR 200 mg Film Tablet; Drug: AVIGAN 200 mg Film Tablets

INTERVENTIONS:
Drug: FAVICOVIR 200 mg Film Tablet — FAVICOVIR 200 MG FT is containing 200 mg favipiravir manufactured by Atabay, Turkey.
  Other Names: Favipiravir 200 MG FT
Drug: AVIGAN 200 mg Film Tablets — AVIGAN 200 mg FT is containing 200 mg favipiravir manufactured by Toyama, Japan.
  Other Names: Favipiravir 200 mg FT

SUMMARY:
A single dose of Reference product containing 200 mg favipiravir and a single dose of Test product containing 200 mg favipiravir or vice versa; administered with 240 mL of water at room temperature, in each period under fasting conditions with current pandemic precautions.

DETAILED DESCRIPTION:
Favipiravir is a drug with a mechanism of action different from that of the existing influenza antiviral drugs and effective against all types and sub-types of human influenza A, B and C viruses in vitro, showing anti-viral activity against various influenza virus strains including avian and swine viruses. Favipiravir also has shown anti-viral activity even against amantadine, oseltamivir and zanamivir-resistant influenza viruses in vitro. The mechanism of action of favipiravir is the selective inhibition of RNA polymerase by favipiravir ribosyl triphosphate formed by cellular enzymes in the influenza virus leading to antiviral activity.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian male subjects aged between 20 and 40 years
2. Non smokers or smoking maximum 5 cigarettes a day, those who won't smoke or drink coffee during the study period
3. Two Negative Covid-19 PCR test results
4. Negative alcohol breath test results
5. Normal physical examination at screening visit
6. Having the Body Mass Index ranged between 18.5-30 kg/m2 (see Appendix I) which is in the desirable range according to the age
7. Ability to communicate adequately with the investigator himself or his representatives
8. Ability and agreement to comply with the study requirements
9. Normal blood pressure and heart rate measured under stabilised conditions at the screening visit after at least 5 minutes of rest under supine position: SBP within 100 to 140 mmHg, DBP within 60 to 90 mmHg and HR within 50 to 90 bpm
10. Normal/ acceptable 12-lead electrocardiographic results at least after 5 minutes of rest
11. Laboratory results within normal range or clinically non-significant (CBC, glucose, urea, uric acid, creatinine, estimated GFR (eGFR), total bilirubin, sodium, potassium, calcium, chloride, SGOT (AST), SGPT (ALT), GGT, alkaline phosphatase, total protein and urinalysis), drug addiction scanning in urine results in negative (amphetamine, barbiturate, benzodiazepine, cannabinoid, cocaine, opiate)
12. Understanding of the study and agreement to give a written informed consent according to section 20.3
13. Understanding of that he and his partner will use a practice adequate contraception during the study and at least 7 days after the study
14. Volunteer's compliance with isolation rules defined at study protocol

Exclusion Criteria:

1. Who have atopic constitution or asthma or known allergy for favipiravir and/or any other ingredients of the products.
2. Any history or presence of clinical relevance of cardiovascular, neurological, musculoskeletal, haematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolism or psychiatric disease, any type of porphyria.
3. Symptomatic or asymptomatic orthostatic hypotension at screening or before the first drug administration defined by a decrease of SBP more than 20 mmHg or DBD more than 10 mmHg occurs between sitting/supine to standing position subject will be excluded (if it deemed necessary by the investigator),
4. Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or except herniotomy.
5. Subjects who have given more than 400 mL blood within the last two months before the first drug administration and subjects who have participated to any drug research within the last two months before the first drug administration.
6. Subjects suspected to have a high probability of non-compliance to the study procedure and/or completion of the study according to the investigator's judgement.
7. Subjects who used any of prescribed systemic or topical medication (including OTC medication) within 2 weeks (or six elimination half lives of this medication, whichever is longer) before the initiation of the study (except single doses of analgesics which have no drug interaction with study product).
8. Use of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
9. History of allergic response to heparin.
10. Subjects who have any chronic disease which might interfere with absorption, distribution, metabolism or excretion of the drug.
11. Subjects who regular consumed of beverages or food containing methylxanthines (e.g. coffee, tea, cola, caffeine, chocolate, sodas,) equivalent to more than 500 mg methylxanthines per day.
12. Subjects who has taken any grapefruit or grapefruit juice during 7 days prior to drug administration, during the study.
13. History of drug abuse.
14. History of alcohol abuse and/or regular use of more than 2 units of alcohol per day or 10 units per week and/or positive alcohol breath test results (Note: one unit of alcohol equals 250 mL beer, 125 mL wine or 25 mL spirits).
15. Positive blood test for HBV, HCV and HIV.
16. Who have relationship to the investigator.
17. Who are not suitable to any of inclusion criteria.
18. History of difficulty of swallowing.
19. Intake of depot injectable solutions (including study medications) within 6 months before start of the study.
20. Intake of enzyme-inducing, organotoxic or long half-life drugs within 4 weeks before start of the study.
21. Special diet due to any reason, e.g. vegetarian.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muradiye Nacak, MD,PhD, Principal Investigator — Farmagen Ar-Ge Biyot. Ltd. Sti
Locations (2):
- Turkey (Türkiye) (2):
  - Novagenix Drug R&D Center, Akyurt, Ankara
  - Farmagen Ar-Ge Biyot. Ltd. Sti., Şahinbey, Gaziantep

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 57 subject screened
Groups:
- Experimental: FAVICOVIR Then AVIGAN: Participants first received Favicovir 200 mg FT manufactured by Atabay in a fasting state. After a washout period of 48 hours, they then received Avigan FT200 mg manufactured by Toyama Chemical Industry Co.Ltd./Japan in a fasting state.
Period: Period 1
Arm/Group | Experimental: FAVICOVIR Then AVIGAN | AVIGAN Then FAVICOVIR
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Experimental: FAVICOVIR Then AVIGAN | AVIGAN Then FAVICOVIR
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FAVICOVIR Then AVIGAN | AVIGAN Then FAVICOVIR | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Full Range); unit: years] | 29 [25 to 35] | 29 [25 to 35] | 29 [25 to 35]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 15 | 15 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Race/Ethnicity, Customized [Number; unit: subjects]
  Caucasian | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tlast of Favipiravir
Description: Area under the concentration-time curve of favipiravir in plasma over the time interval from 0 to 24 hours
Time Frame: 0 to 24 hours post-dose
Population: 29 subjects were analysed and included in statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Favicovir 200 mg FT: Participants received single oral dose of 200 mg favipiravir (Favicovir 200 mg FT, Atabay-Turkey) under fasting conditions.
- Avigan 200 mg FT: Participants received single oral dose of 200 mg favipiravir (Avigan 200 mg FT, Toyama-Japan) under fasting conditions.
Arm/Group | Favicovir 200 mg FT | Avigan 200 mg FT
Number analyzed (Participants) | 29 | 29
ng*hr/mL | 9641.989 (2545.1) | 9907.170 (2423.5)
Statistical Analysis 1: Comparison: Favicovir 200 mg FT vs Avigan 200 mg FT; Test type: Equivalence — 0.80-1.25 margins for equivalence; p = 0.0000, ANOVA; Mean Ratio = 0.9684, 90% CI 2-sided [0.9400 to 0.9977]

2. Primary Outcome: Cmax of Favipiravir
Description: Maximum plasma concentration of favipiravir
Time Frame: 0 to 24 hours post-dose
Population: 29 subjects were analysed and included in statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Favicovir 200 mg FT | Avigan 200 mg FT
Number analyzed (Participants) | 29 | 29
ng/mL | 5411.624 (2025.6) | 5002.171 (1231.1)
Statistical Analysis 1: Comparison: Favicovir 200 mg FT vs Avigan 200 mg FT; Test type: Equivalence — 0.80 - 1.25 equivalence margin is required; p = 0.0155, ANOVA; Mean Ratio = 1.0555, 90% CI 2-sided [0.9292 to 1.1989]

3. Secondary Outcome: AUC0-inf of Favipiravir
Description: Area under the plasma concentration curve to infinite time of favipiravir
Time Frame: 0 to 24 hours post-dose
Population: 29 subjects were analysed and included in statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Favicovir 200 mg FT | Avigan 200 mg FT
Number analyzed (Participants) | 29 | 29
ng*hr/mL | 9910.494 (2618.9) | 10152.115 (2507.694)
Statistical Analysis 1: Comparison: Favicovir 200 mg FT vs Avigan 200 mg FT; Test type: Equivalence — 0.80 - 1.25 equivalence margin is not required; p = 0.0000, ANOVA; Mean Ratio = 0.9719, 90% CI 2-sided [0.9440 to 1.0006]

4. Secondary Outcome: Tmax of Favipiravir
Description: Time to reach maximum plasma concentration of favipiravir
Time Frame: 0 to 24 hours post-dose
Population: 29 subjects were analysed and included in statistical analysis.
Measure: Mean (Standard Deviation); unit: hr
Groups:
- Favicovir 200 mg FT: Participants received single dose of 200 mg Favipiravir (Favicovir 200 mg FT, Atabay-Turkey) under fasting conditions.
Arm/Group | Favicovir 200 mg FT | Avigan 200 mg FT
Number analyzed (Participants) | 29 | 29
hr | 0.609 (0.343) | 0.733 (0.478)

ADVERSE EVENTS:
Time Frame: 9 days
Groups:
- FAVICOVIR 200 MG FT (Atabay-Turkey): Participants received single oral dose of 200 favipiravir of Atabay-Turkey under fasting conditions.
- AVIGAN 200 MG FT (Toyama-Japan): Participants received single oral dose of 200 favipiravir of Toyama-Japan under fasting conditions.
Arm/Group | FAVICOVIR 200 MG FT (Atabay-Turkey) | AVIGAN 200 MG FT (Toyama-Japan)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT04406194/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT04406194/ICF_001.pdf